CLINICAL TRIAL: NCT05808010
Title: Clinical Study of Umbilical Cord Blood Mononuclear Cell Therapy for the Treatment of Chronic Atrophic Gastritis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Xu Hongwei, Chief Physician, Shandong Provincial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWYX:NO.2022-1037
Record Dates: First submitted 2023-03-17; First posted 2023-04-11 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Chronic Atrophic Gastritis
MeSH Terms: conditions — Gastritis, Atrophic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mononuclear cells+Weifuchun+Hydrotalcite/L-Glutamine and Sodium Gualenate Granules (Experimental)
  Interventions: Biological: Mononuclear cells; Drug: Weifuchun+Hydrotalcite/L-Glutamine and Sodium Gualenate Granules
- Mononuclear cells (Experimental): Mononuclear cells are obtained from umbilical cord blood by density gradient centrifugation
  Interventions: Biological: Mononuclear cells
- Weifuchun+Hydrotalcite/L-Glutamine and Sodium Gualenate Granules (Active Comparator): Weifuchun is a kind of edible Chinese herbal prescription
  Interventions: Drug: Weifuchun+Hydrotalcite/L-Glutamine and Sodium Gualenate Granules

INTERVENTIONS:
Biological: Mononuclear cells — 2 times gastric submucosal injection of mononuclear cells (10^8) at 1 month interval
  Arms: Mononuclear cells; Mononuclear cells+Weifuchun+Hydrotalcite/L-Glutamine and Sodium Gualenate Granules
Drug: Weifuchun+Hydrotalcite/L-Glutamine and Sodium Gualenate Granules — Orally delivered tablets for 7 months. Take it according to the instructions.
  Arms: Mononuclear cells+Weifuchun+Hydrotalcite/L-Glutamine and Sodium Gualenate Granules; Weifuchun+Hydrotalcite/L-Glutamine and Sodium Gualenate Granules

SUMMARY:
To evaluate the efficacy and safety of umbilical cord blood mononuclear cells in the treatment of chronic atrophic gastritis.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participated in the study and signed an informed consent.
2. The age is 18-65 years old, regardless of gender.
3. Patients with chronic atrophic gastritis by gastroscopy and pathological examination.
4. Patients with a negative C13 breath test or have eradicated Helicobacter pylori infection.
5. Patients without contraindications to submucosal injection of umbilical cord blood derived mononuclear cells.

Exclusion Criteria:

1. Patients with gastric ulcer, erosive gastritis, active upper gastrointestinal bleeding, gastric varices, or other gastric tumors.
2. Patients who are taking or have taken proton pump inhibitors, antibiotics, glucocorticoids, nonsteroidal anti-inflammatory drugs and immunosuppressants in the last six months.
3. People who have had gastric surgery or required gastric surgery during the study.
4. Patients with severe systemic diseases (diseases of cardiovascular, liver, blood, kidneys, lungs or liver).
5. Pregnant or nursing females.
6. Patients who are reluctant to accept endoscopy and treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline OLGA/OLGIM stages of gastric mucosa | At the first, seventh and thirteenth month of treatment
  Assessment of OLGA/OLGIM stages by GI pathologists. The obtained biopsy specimens will be scored using visual analogue scale (0, 1, 2, 3 points for none, mild, moderate and severe, respectively) to evaluate gastroatrophy and gastrointestinal metaplasia
Change from baseline gastric mucosal status under gastroscope | At the first, seventh and thirteenth month of treatment
  Assessment of Kimura-Takemoto classification by endoscopy. The variation of atrophy can reflect the extent and degree of atrophy. The severity of atrophy increases gradually with C1-C2-C3-O1-O2-O3. Cases of closed-type gastric mucosa atrophy have an atrophic boundary between the fundic mucosa and the pyloric mucosa in the antrum or less curvature of the gastric body. Cases of open-type gastric mucosa atrophy have an atrophic boundary in the lateral wall or greater curvature of the gastric body. C, closed; O, open

SECONDARY OUTCOMES:
Change from baseline blood test result | At the first, seventh and thirteenth month of treatment
  Assessment of Gastrin-17 and Pepsinogen I/II
Incidence of adverse reactions | Through follow-up period completion, an average of 1 year
  Assessment of incidence of adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: hongwei Xu, MD, Principal Investigator — Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China